CLINICAL TRIAL: NCT04297111
Title: Effect of Bacillus Coagulans on Skeletal Muscle Protein Synthesis in Response to Vegetable Protein Ingestion
Brief Title: Probiotic-Muscle Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College Dublin (Other)
Collaborators: Kerry Group (Unknown)
Responsible Party: Principal Investigator, Prof Helen M Roche, Professor Helen Roche, University College Dublin
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: IRCEB
Record Dates: First submitted 2020-03-03; First posted 2020-03-05 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Old Age; Debility; Muscle Weakness; Protein Deregulation; Protein Deposition
MeSH Terms: conditions — Frailty; Muscle Weakness | interventions — Probiotics

STUDY DESIGN:
Intervention Model Description: The study will be a randomised, double-blind, placebo-controlled crossover study. Each participant will undergo 8 weeks of Bacillus coagulans (probiotic) supplementation and 8 weeks of placebo supplementation in a counterbalanced order. There will be a 5-day trial period at the end of each supplementation phase. There will be a wash-out period of 8 weeks between probiotic and placebo supplementation.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Maltodextrin containing capsule
  Interventions: Other: Placebo
- Probiotic (Experimental): Probiotic containing capsule
  Interventions: Dietary Supplement: Probiotic

INTERVENTIONS:
Dietary Supplement: Probiotic — GanedenBC30 (Bacillus coagulans GBI-30, 6086) capsule made of 1 billion colony forming units (cfu). Description: pure cell mass of an L-(+) lactic acid-producing, gram-positive, spore-forming shaped bacterium that is aerobic to microaerophilic. Maltodextrin used as filler.
  Arms: Probiotic
Other: Placebo — Maltodextrin capsule, no active ingredient
  Arms: Placebo

SUMMARY:
This study will examine the effect of probiotic supplementation (Bacillus coagulans) on muscle protein synthesis in older adults in response to a plant-based diet.

The investigators hypothesize that probiotic supplementation will enhance the digestibility of plant protein, therefore increasing the proportion of ingested amino acids that appear in systemic circulation and enhancing rates of muscle protein synthesis.

DETAILED DESCRIPTION:
There is increasing interest in the use of plant-based proteins, both from the perspectives of global sustainability and growing consumer markets; however, plant-based proteins are known to have lower digestibility and lower ability to stimulate muscle protein synthesis (an important determinant of muscle mass) compared with animal-based proteins. Emerging evidence indicates that the probiotic Bacillus coagulans GBI-30, 6086 (GanedenBC30) can enhance plant protein digestibility. As such, Bacillus coagulans treatment may augment rates of muscle protein synthesis in response to plant-based protein intake in humans, by increasing the proportion of ingested amino acids that appear in systemic circulation after a plant meal, as circulating amino acids act as both a trigger to stimulate muscle protein synthesis in humans as well as providing the building block for new muscle tissue. An increase in muscle protein synthesis rates would be particularly critical in older adults as it is well established that one of the key mechanisms driving the loss of muscle mass with age is a reduction in muscle protein synthesis rates in response to dietary protein intake. Therefore, if probiotic supplementation can improve muscle protein synthesis rates following plant protein consumption, this indicates it may represent an effective and environmentally sensitive strategy to attenuate adverse age-related loss of muscle mass and muscle function. This is critical as the maintenance of skeletal muscle health is an important factor in the preservation of independence and quality of life as we age.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥65 y
* Sex: males and female
* Body mass index (BMI) between 20-35 kg/m2
* Non-smokers
* Generally healthy according to responses to a standard health screening questionnaire

Exclusion Criteria:

* Cancer (malignancy in the past 5 years)
* CVD
* Chronic kidney disease
* Liver failure
* Diabetes or pre-diabetes
* Conditions that will affect the ability to consume, digest and/or absorb the study supplement (i.e. gastrointestinal disease)
* Smokers
* Excess alcohol intake
* Regular resistance training
* Total walking incapacity
* Musculoskeletal or neuromuscular impairments
* Medications interfering with muscle metabolism
* Ongoing probiotic supplementation
* Antibiotic use in the previous 6 weeks
* Significant body mass loss in the 1 month period prior to the study

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-11-25 (Actual); Primary Completion 2020-10-03 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Myofibrillar protein synthesis | 6 months
  Measured as fractional synthetic rate (%/day) over a 2-d period after each supplementation arm and in response to a plant-based diet
Pattern of change in plasma total amino acid, essential amino acid and leucine concentrations | 6 months
  Assessed via GC-MS.

SECONDARY OUTCOMES:
Changes in microbiome composition | 6 months
  Assessed in faecal samples via 16s rRNA analysis
Change in metabolome | 6 months
  Assesed in blood and faecal water via 600 MHz nuclear magnetic resonance (NMR) spectrometry
Changes in gut hormones | 6 months
  ELISA (enzyme-linked immunosorbent assay)
Changes in gut/digestion-related complaints | 6 months
  Assessed via the Gastrointestinal Symptom Rating Scale (GSRS), where minimum and maximum values are: no discomfort at all, and very severe discomfort respectively (higher score means worse outcome).
Changes in bowel movement | 6 months
  Assessed via the Bristol Stool chart, where average faecal appearance is indicated out of seven options available
Changes in strength | 6 months
  Assessed via handgrip strength using a handgrip dynamometer
Changes in immuno-surveillance | 6 months
  Assessed via the Common Cold Questonnaire (CCQ), where minimum and maximum values are: none, and severe respectively (higher score means worse outcome).
Changes in appetite | 6 months
  Assessed via the Visual Analogue Scale (VAS) during 3 days of the trial period and after the protein-containing beverage, where the left and right side of the scale indicate: not hungry at all, and extremely hungry respectively (there is not an assigned better or worse outcome for this scale)

CONTACTS AND LOCATIONS:
Overall Officials: Helen Roche, PhD, Principal Investigator — University College Dublin; Caoielann Murphy, PhD, Study Director — University College Dublin
Locations (1):
- University College Dublin, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No
Research results will be published in a peer-reviewed journal once the study has finalised and the data has been analized.